CLINICAL TRIAL: NCT02900989
Title: Etude de Validation de la Version française d'un Questionnaire " Ask Suicide-Screening Questions " (ASQ) Dans Une Population de Patients Adolescents Pris en Charge en unité d'Urgences pédiatriques
Brief Title: Validation of the French Version of Ask Suicide-Screening Questions (ASQ) in Adolescents Managed in Pediatric Emergency Unit
Acronym: ASQ-Fr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2016/CHU/01
Record Dates: First submitted 2016-09-06; First posted 2016-09-15 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Suicidal Ideation
Keywords: Psychiatry; Pediatrics; Suicide
MeSH Terms: conditions — Suicidal Ideation; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASQ-Fr (Other): Adolescents undergo the ASQ-Fr questionnaire composed of 5 items.
  Interventions: Behavioral: Suicide screening
- SIQ-Fr (Other): Adolescents undergo the SIQ-Fr questionnaire composed of 30 items if >=15 yo and the SIQ-Fr Junior composed of 15 items if <15 yo
  Interventions: Behavioral: Suicide screening

INTERVENTIONS:
Behavioral: Suicide screening — Patients of the emergency unit usually do not pass this kind of questionnaire in the absence of warning signs. Then it could result in adverse effects on behavior and ideation.
  The study had to be declared as an interventional study according to French law.

SUMMARY:
The ASQ-Fr study aims at validating the French version of Ask Suicide-Screening Questions composed of 5 items in adolescents managed in pediatric emergency department. Therefore, use of this brief valid screening instrument could assess the risk for suicide in pediatric patients and then improve the prevention of suicidal tendencies in this population.

DETAILED DESCRIPTION:
ASQ-Fr is a prospective, cross-sectional instrument-validation study evaluated 5 candidate screening questions assessing suicide risk in adolescents between 10 and 18 years of age managed in two urban, pediatric emergency departments associated with tertiary care hospitals.

ASQ-Fr questionnaire is conducted by a psychologist before or after the French version of the SIQ/SIQ Junior (Suicidal Ideation Questionnaire), depending on the randomisation in the unit. SIQ is composed of 30 items and valid for adolescents aged 15 years or more. SIQ Junior is composed of 15 items and valid for children up to 14 years old.

Questionnaires are followed by an interview in adolescents and parents separately by the psychologist to evaluate perceptions, feasibility and acceptability of questionnaires.

It is planned a convenience sample of 200 patients aged 10 to 18 years who presented with either medical or surgical chief concerns to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* patient with informed consent of adolescents and at least one of parents or a guardian
* patient with social protection cover
* in adequation with emergency management

Exclusion Criteria:

* patients with mental disorder
* minor without parent/gardian at the emergency unit

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Proportion of adolescents detected at suicide risk by the French version of Ask Suicide-Screening Questions and by the SIQ or SIQ Junior | 6 months
  Adolescents are interviewed by the psychologist who administer SIQ/SIQ Junior questionnaire then ASQ or the opposite according to the randomisation process

SECONDARY OUTCOMES:
Type and proportion of answers about perceptions by parents of a questionnaire on suicidal ideation conducted in their child | 6 months
  Questionnaires are followed by an interview in adolescents and parents separately by the psychologist
Type and proportion of answers about perceptions by adolescent of the questionnaires | 6 months
  Questionnaires are followed by an interview in adolescents and parents separately by the psychologist

CONTACTS AND LOCATIONS:
Overall Officials: Erick Gokalsing, MD, Study Director — INSERM U1178
Locations (1):
- Centre Hospitalier Universitaire de La Réunion, Saint-Pierre, France